CLINICAL TRIAL: NCT03378336
Title: Psoriatic Arthritis Research Collaborative: Biologic Sub-Study
Acronym: PARC-B
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: The Cleveland Clinic (Other); NYU Langone Health (Other); University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: 828357
Record Dates: First submitted 2017-11-27; First posted 2017-12-19 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Approximately 40 mL (4 tubes) of blood will be drawn at each of 2 visits. The blood and information collected throughout this study will be used to build a repository for future research projects. The de-identified information stored in the redcap will available only to the study teams at each of the sites involved in this study and to those PIs for future research. Blood samples will be processed and stored at individual sites. De-identified blood samples may be shipped to a central location for further testing on bio-markers of treatment response and disease progression.
  Participants may retract permission and ask that their samples be destroyed. Information from these samples is exploratory and will not be shared with participants or included in medical records
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Group: This is an observational study with only one group/cohort with no intervention

SUMMARY:
Psoriatic arthritis (PsA) is an inflammatory arthritis with substantial variation in clinical features. We propose a multicenter collaborative approach to better understand the phenotypes and current management of PsA in the United States.The central goal of this proposal is to obtain the data necessary to design a pragmatic trial in PsA.

DETAILED DESCRIPTION:
Psoriatic arthritis (PsA) is a chronic inflammatory arthritis that can be associated with devastating outcomes including irreversible joint damage. The management of a patient with PsA is extremely challenging due to the high degree of phenotypic heterogeneity. The ultimate goal of this proposal is to prepare pragmatic trials in PsA trials that will encompass all relevant subgroups of patients. The aims of this study specifically focus on responses to biologic therapy among patients with PsA and determining the optimal set of outcome measures for PsA trials.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-89
* Active PsA (at least one swollen joint or enthesitis) -Meet CASPAR criteria (Table 2) (103) -Initiation of TNFi (etanercept, adalimumab, infliximab, certolizumab, golimumab) (At the time of the submission, TNFi biosimilars have been approved by the FDA but are not available on the US market. Once available, patients starting TNFi biosimilars will similarly be eligible for participation. Patients may have been on the medication in the past but must have had greater than 2 months off the medication.Patients may be taking other traditional DMARDs. A washout period is not required.)

Exclusion Criteria:

* Unable to give informed consent
* Out of the age range
* Switching therapies for skin psoriasis in the setting of well controlled joint and enthesis symptoms.
* Patients with only active PsA

Ages: 18 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Rheumatology clinic patients with active PsA switching to or adding a TNFi.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2017-12-31 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Ogdie, MD, Principal Investigator — University of Pennsylvania
Locations (4):
- United States (4):
  - NYU School of Medicine, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Hospital at the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
All four institutions use the Epic electronic medical record system and have existing REDCap databases. For the purpose of this study and use in future studies, we will build a PARC Core REDCap Database. All four institutions will have access to this Core REDCap Database with designated data use agreements. The PARC Core REDCap Database will then be populated from each of our existing institutional RedCap databases. Personal identifiers (name, medical record number) will not be stored as a part of this dataset. Instead, personal identifiers will remain within each individual institution and only de-identified data placed in the Core REDCap database. To ensure the protection of the subjects and data integrity, we will maintain the highest security settings for the Core REDCap Database.
Supporting Information: SAP, ICF
Time Frame: This data will be accessible throughout and after completion of the study.
Access Criteria: The de-identified information stored in the redcap will available only to the study teams at each of the sites involved in this study and to those PIs for future research. Researchers not involved in this study will not be permitted to request or use data or samples from this study.

REFERENCES:
- [Derived] Reddy SM, Xue K, Husni ME, Scher JU, Stephens-Shields AJ, Goel N, Koplin J, Craig ET, Walsh JA, Ogdie A. Use of the Bath Ankylosing Spondylitis Disease Activity Index in Patients With Psoriatic Arthritis With and Without Axial Disease. J Rheumatol. 2024 Feb 1;51(2):139-143. doi: 10.3899/jrheum.2023-0504. PMID 38101918
- See also: Responsiveness and Minimum Clinically Important Difference in Patient-Reported Outcome Measures Among Patients With Psoriatic Arthritis: A Prospective Cohort Study — https://pubmed.ncbi.nlm.nih.gov/36913210/
- See also: Use of the Bath Ankylosing Spondylitis Disease Activity Index in Patients With Psoriatic Arthritis With and Without Axial Disease — https://pubmed.ncbi.nlm.nih.gov/38101918/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 171 unique participants were enrolled in the study, but there were 266 instances of treatment initiation analyzed (each participant could initiate >1 therapy).
  Of the 266 instances of treatment initiation, not all outcome measures were completed at both Baseline and Month 3. Therefore, some outcome measures have a smaller number of units analyzed to include only those completed at both timepoints.
Units Other Than Participants: Treatment Initiations
Groups:
- Participants With PsA Starting a New Therapy: This is an observational study with only one group - participants with PsA starting a new therapy.
Period: Overall Study
Arm/Group | Participants With PsA Starting a New Therapy
Started | 171; 266 Treatment Initiations
Completed | 171; 266 Treatment Initiations
Not Completed | 0; 0 Treatment Initiations

BASELINE CHARACTERISTICS:
Population: Among the 171 unique participants, there were 266 instances of treatment initiation analyzed (each participant could initiate >1 therapy)
Units Other Than Participants: treatment initiations
Arm/Group | Observational Group
Number analyzed (Participants) | 171
Number analyzed (treatment initiations) | 266
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (13.8)
Sex: Female, Male [Count of Units; unit: treatment initiations]
  Female | 140
  Male | 126
Ethnicity (NIH/OMB) [Count of Units; unit: treatment initiations]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 229
  Unknown or Not Reported | 17
Race (NIH/OMB) [Count of Units; unit: treatment initiations]
  American Indian or Alaska Native | 4
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 242
  More than one race | 0
  Unknown or Not Reported | 18
Tender joint count [Mean (Standard Deviation); unit: joints] | 5.8 (7.4)
Swollen joint count [Mean (Standard Deviation); unit: joints] | 2.9 (4.9)
Body surface area (%) [Mean (Standard Deviation); unit: %] | 1.6 (3.9)
Enthesitis count [Mean (Standard Deviation); unit: entheses] | 0.6 (1.1)
Dactylitis count [Mean (Standard Deviation); unit: digits] | 0.3 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Patient Function Response to Biologic Therapy as Measured by RAPID3
Description: Patient's perception of response to therapy as related to patient functionality. Measured by a change in RAPID3 score from baseline to 3 month visit.
  RAPID3 (Routine Assessment of Patient Index Data 3) is a pooled index of the 3 patient-reported American College of Rheumatology Core Data Set measures: function, pain, and patient global estimate of status. Each of the 3 individual measures is scored 0 to 10, for a total of 30. Disease severity may be classified on the basis of RAPID3 scores: >12 = high; 6.1-12 = moderate; 3.1-6 = low; < or =3 = remission.
Time Frame: 3 Months
Population: 225 completed RAPID3 at Baseline and Month 3
Measure: Mean (Standard Deviation); unit: change in score
Units Other Than Participants: treatment initiations
Arm/Group | Observational Group
Number analyzed (Participants) | 171
Number analyzed (treatment initiations) | 225
change in score | -1.11 (5.26)

2. Secondary Outcome: Patient Function Response to Biologic Therapy as Measured by HAQ-DI
Description: Patient's perception of response to therapy as related to patient functionality. Measured by change in HAQ-DI score from baseline to 3 month visit.
  The HAQ-DI (Health Assessment Questionnaire - Disability Index) covers 20 items in eight domains related to measuring difficulty in performing activities of daily living. Each question is rated on a 0-3 scale, where 0 indicates "without difficulty" and 3 indicates "unable to do." The highest score in each domain is accepted as the score in that domain. Scores for the 8 domains are averaged to compute final score between 0 and 3. Scores 0-1 indicate mild to moderate disability, 1-2 indicate moderate to severe disability, and 2-3 indicate severe to very severe disability.
Time Frame: 3 Months
Population: 85 participants completed HAQ-DI at Baseline and Month 3
Measure: Mean (Standard Deviation); unit: change in score
Units Other Than Participants: treatment initiations
Arm/Group | Observational Group
Number analyzed (Participants) | 85
Number analyzed (treatment initiations) | 85
change in score | -0.07 (0.42)

3. Secondary Outcome: Patient Quality of Life Response to Biologic Therapy as Measured by PROMIS10
Description: Patient's perception of response to therapy as related to quality of life. Measured by change in PROMIS10 Physical Health score from baseline to 3 month visit.
  PROMIS10 (Patient-Reported Outcomes Measurement Information System) Physical Health is a 10-item questionnaire, each with a five point scale from Poor to Excellent. PROMIS uses Item Response Theory (IRT) statistical model that links individual questions to a presumed underlying trait or concept of global health represented by all items in the scale; instruments are scored using item-level calibrations ("response pattern scoring") in an online tool (T-Score range 0-100). Increasing score indicates improvement.
Time Frame: 3 Months
Population: 183 instances of therapy initiation completed PROMIS10 PH at Baseline and Month 3.
Measure: Mean (Standard Deviation); unit: change in score
Units Other Than Participants: therapy initiation
Arm/Group | Participants With PsA Starting a New Therapy
Number analyzed (Participants) | 171
Number analyzed (therapy initiation) | 183
change in score | 1.43 (6.20)

4. Secondary Outcome: Patient Quality of Life Response to Biologic Therapy as Measured by PSAID
Description: Patient's perception of response to therapy as related to quality of life. Measured by change in PSAID score from baseline to 3 month visit.
  PSAID (PsA Impact of Disease) is a questionnaire composed of 12 health domains, examining different perspectives (both physical and psychological). Each domain is evaluated by a single question with a range from 0-10 in which higher results indicate a greater impact of the disease. Individual domain scores are weighted to indicate those with a greater effect, then the sum of weighted domain scores is divided by 20 to compute the final score (range 0-10).
Time Frame: 3 Months
Population: 225 instances of therapy initiation completed PSAID at Baseline and Month 3.
Measure: Mean (Standard Deviation); unit: change in score
Units Other Than Participants: therapy initiations
Arm/Group | Participants With PsA Starting a New Therapy
Number analyzed (Participants) | 171
Number analyzed (therapy initiations) | 225
change in score | -0.30 (1.05)

5. Secondary Outcome: Physician Assessment of Disease Response to Biologic Therapy as Measured by Swollen Joint Count.
Description: Physician assessment of disease activity as measured by change in swollen joint count from baseline to 3 months.
Time Frame: 3 Months
Population: 256 instances of therapy initiation had swollen joint count measured at Baseline and Month 3
Measure: Mean (Standard Deviation); unit: change in joint count
Units Other Than Participants: therapy initiations
Arm/Group | Participants With PsA Starting a New Therapy
Number analyzed (Participants) | 171
Number analyzed (therapy initiations) | 256
change in joint count | -0.81 (4.71)

6. Secondary Outcome: Physician Assessment of Disease Response to Biologic Therapy as Measured by Tender Joint Count.
Description: Physician assessment of disease activity as measured by change in tender joint count from baseline to 3 months.
Time Frame: 3 Months
Population: 256 instances of therapy initiation had tender joint count measured at Baseline and Month 3.
Measure: Mean (Standard Deviation); unit: change in joint count
Units Other Than Participants: therapy initiations
Arm/Group | Participants With PsA Starting a New Therapy
Number analyzed (Participants) | 171
Number analyzed (therapy initiations) | 256
change in joint count | -0.63 (8.35)

7. Secondary Outcome: Disease Activity and Response to Biologic Therapy as Measured by Patient Pain Assessment
Description: Disease Activity and Response to Biologic Therapy as measured by change in Patient Pain Assessment from baseline to 3 month visit.
  The Patient Pain Assessment is measured on a scale of 0-100 where a higher score indicates worse pain.
Time Frame: 3 Months
Population: 234 instances of therapy initiation completed the Pt Pain assessment at Baseline and Month 3.
Measure: Mean (Standard Deviation); unit: change of score
Units Other Than Participants: therapy initiations
Arm/Group | Participants With PsA Starting a New Therapy
Number analyzed (Participants) | 171
Number analyzed (therapy initiations) | 234
change of score | -0.75 (2.66)

8. Secondary Outcome: Disease Activity and Response to Biologic Therapy as Measured by Physician Global Assessment
Description: Disease Activity and Response to Biologic Therapy as measured by change in Physician Global Assessment from baseline to 3 month visit.
  Physician Global Assessment is measured on a scale from 0-10 where a higher score indicates greater disease impact.
Time Frame: 3 Months
Population: 249 instances of therapy initiation had a Physician Global Assessment at Baseline and Month 3.
Measure: Mean (Standard Deviation); unit: change in score
Units Other Than Participants: therapy initiations
Arm/Group | Participants With PsA Starting a New Therapy
Number analyzed (Participants) | 171
Number analyzed (therapy initiations) | 249
change in score | -0.30 (1.54)

9. Secondary Outcome: Disease Activity and Response to Biologic Therapy as Measured by Patient Global Assessment
Description: Disease Activity and Response to Biologic Therapy as measured by change in Patient Global Assessment from baseline to 3 month visit.
  Patient Global Assessment is measured on a scale of 0-10 where a higher score indicates greater disease impact.
Time Frame: 3 Months
Population: 234 instances of therapy initiation completed the Pt Global assessment at Baseline and Month 3.
Measure: Mean (Standard Deviation); unit: change in score
Units Other Than Participants: therapy initiations
Arm/Group | Participants With PsA Starting a New Therapy
Number analyzed (Participants) | 171
Number analyzed (therapy initiations) | 234
change in score | -0.24 (2.66)

ADVERSE EVENTS:
Time Frame: AE data were collected for each participant for 1 year.
Arm/Group | Observational Group
All-Cause Mortality (participants affected / at risk) | 0/171
Serious Adverse Events (participants affected / at risk) | 0/171
Other Adverse Events (participants affected / at risk) | 0/171

LIMITATIONS AND CAVEATS:
171 unique participants were enrolled in the study, but there were 266 instances of treatment initiation analyzed (each participant could initiate >1 therapy).

Of the 266 instances of treatment initiation, not all outcome measures were completed at both Baseline and Month 3. Therefore, some outcome measures have a smaller number of units analyzed to include only those completed at both timepoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-14): https://cdn.clinicaltrials.gov/large-docs/36/NCT03378336/Prot_SAP_000.pdf